CLINICAL TRIAL: NCT07292233
Title: A Randomized, Open-Label, Single-Dose, Two-Period, Crossover Phase I Clinical Study to Evaluate the Food Effect on the Pharmacokinetics of LPM787000048 Maleate Extended-Release Tablets (LY03020) in Healthy Subjects
Brief Title: A Food Effect Study of LY03020 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03020/CT-CHN-102
Record Dates: First submitted 2025-08-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Alzheimer's Disease Psychosis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- fasted,fed (Experimental): Subjects will take LY03020 80mg under fasted conditions and after a standard high-fat breakfast in period 1 and 2 respectively.
  Interventions: Drug: LY03020
- fed,fasted (Experimental): Subjects will take LY03020 80mg after a standard high-fat breakfast and under fasted conditions in period 1 and 2 respectively.
  Interventions: Drug: LY03020

INTERVENTIONS:
Drug: LY03020 — single dose，administered orally for each period

SUMMARY:
This is a randomized, open-label, single-dose, two-period, crossover study to assess the food effect on pharmacokinetics (PK) and safety of LY03020 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign informed consent voluntarily.
* Male or female aged 18 to 45 years.
* Body weight ≥ 50.0kg for male and ≥ 45.0kg for female, and body mass index (BMI) between 18.5 and 26.0 kg/m2.

Exclusion Criteria:

* Subjects have any clinically significant medical condition or chronic disease.
* Subjects experienced a history of keratopathy, fundus disease, increased intraocular pressure, or angle-closure glaucoma. Subjects have any abnormal and clinically significant test for ophthalmic examination during screening.
* Subjects with a history of orthostatic hypotension or syncope.
* Subjects with condition that may interfere with the drug absorption, distribution, metabolism and excretion significantly.
* Subjects had a history of surgery within 3 months prior to administration, or had not recovered, or have a surgical plan during the study.
* Subjects have any clinically significant abnormal vital signs, laboratory values, and ECGs.
* Subjects have used any of nonprescription drugs within 7 days or prescription drugs within 28 days prior to first dosing.
* Subjects have a history of allergic diseases, or allergic to any substance contained in the formulation.
* Subjects have a positive test for HBsAg, HCV-Ab, HIV-Ab, or syphilis antibody.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of LPM787000048 in plasma | up to Day 12
Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of LPM787000048 in plasma | up to Day 12
Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC0-t) of LPM787000048 in plasma | up to Day 12

SECONDARY OUTCOMES:
Time to maximum observed concentration (Tmax) of LPM787000048 in plasma | up to Day 12
Apparent terminal elimination half-life (t1/2) of LPM787000048 in plasma | up to Day 12
Number of participants with adverse events (AEs). | up to Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing AnDing Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No